CLINICAL TRIAL: NCT02003092
Title: A Multi-Center, Dose Finding, Open Label, Phase 1 Study of RX-5902 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: RX-5902 Treatment of Subjects With Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rexahn Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RX-5902-P1-01
Record Dates: First submitted 2013-11-15; First posted 2013-12-06 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumor; Triple Negative Breast Cancer
Keywords: Metastatic; Rexahn; Phase 1; Triple Negative Breast Cancer; Phase 2; Relapsed
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis; Recurrence | interventions — RX-5902

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RX-5902 (Experimental): RX-5902 will be taken daily for 4 weeks in each 4 week cycle. Subjects will be fasting for 8 hours before and food may be ingested approximately 3 hours after the dose has been administered.
  Interventions: Drug: RX-5902

INTERVENTIONS:
Drug: RX-5902 — escalating doses (mg)
  Other Names: Supinoxin™

SUMMARY:
The purpose of this Phase 2 portion of the study is to use the dose and schedule of RX-5902 identified in the phase 1 to treat subjects with triple negative breast cancer.

DETAILED DESCRIPTION:
In this dose-finding, open-label, single-agent study of RX-5902, subjects will be treated for up to 6 cycles of therapy. RX-5902 will be administered orally daily for 3 weeks followed by 1 week of rest in each cycle. All subjects will be followed for at least 30 days after the last dose of study agent for safety.

ELIGIBILITY:
Inclusion Criteria:

* Male and female who are 18 yrs or older
* Histologically confirmed triple negative breast cancer that are refractory, intolerant, or ineligible to receive approved standard therapies
* Measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST)
* Life expectancy of at least 3 months
* Able to swallow capsules
* Provide written informed consent

Exclusion Criteria:

* Primary brain tumor or active brain metastasis
* Not recovered to less than or equal to Grade 1 toxicities (except Grade 2 alopecia or neuropathy) associated with previous cancer therapies
* Any other cancer treatments within 2 weeks of planned study treatment
* History of any medical or psychiatric condition or addictive disorder, or lab abnormality that in the opinion of the investigator, may increase risks or may interfere with study participation or interpretation of study results
* History of clinically significant GI bleed, intestinal obstruction, or GI perforation within 6 months of study dose
* Uncontrolled diabetes
* History of long QT syndrome or clinically significant cardiac arrhythmias (except stable atrial fibrillation)
* Myocardial infarction within 6 months of study dose
* Active infection requiring IV antibiotics within 2 weeks of study dose
* History of Hepatitis B, C, or HIV
* Use of potent inhibitor or inducer of CYP3A4/3A5 within 14 days of planned study treatment or expected requirement for use of such a drug during study
* Use of a potent inhibitor or inducer of drug transporters or conjugating enzymes within 14 days prior to planned study treatment or expected requirement for use of such a drug during study
* Receiving other investigational agents or not yet completed 30 days since completion of an investigational study
* Pregnant, planning a pregnancy, or breast feeding
* Male or female not willing to use adequate contraceptive precautions during the study period. Females must either be surgically sterile, post-menopausal for 12 months, or use a contraceptive approved by sponsor.
* Unwilling or unable to provide written informed consent, comply with study requirements, or be available for follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2019-10 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) (Phase 1) | after 4 weeks of treatment with RX-5902
Progression free survival rate and/or overall clinical response rate (Phase 2) | 16 weeks of treatment with RX-5902

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of RX-5902 | predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8 hrs after the first dose
Changes in tumor size mm | baseline and 24 weeks
Time to progression (Phase 2) | Baseline and at 4, 8, 12, 16 and 24 weeks
Duration of response (Phase 2) | Baseline and at 4, 8, 12, 16 and 24 weeks
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months

OTHER OUTCOMES:
phosphorylated P68 by IHC | baseline and 8 weeks
Tumor burden response (Phase 2) | Baseline and at 4, 8, 12, 16 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ely Benaim, MD, Study Director — Rexahn Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - Rexahn site, Tucson, Arizona
  - Rexahn Site, Aurora, Colorado
  - Rexahn site, Chicago, Illinois
  - Rexahn Site, Detroit, Michigan
  - Rexahn Site, Hackensack, New Jersey
  - Rexahn Site, New York, New York
  - Rexahn Site, Greenville, South Carolina
  - Rexahn site, Arlington, Virginia